CLINICAL TRIAL: NCT00877695
Title: Young Hispanic Men "Entre Culturas": Navigating Culture, Identity and HIV Risk
Brief Title: Motiv82Change: an HIV Prevention Study for Young Latino Men
Acronym: Motiv82Change
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: Entre Culturas
Record Dates: First submitted 2009-04-06; First posted 2009-04-08 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-02

CONDITIONS: HIV Infections
Keywords: HIV; HIV Seronegativity; prevention; Hispanic; Latino; MSM; men
MeSH Terms: conditions — HIV Infections; Multiple Endocrine Neoplasia Type 1

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Motive8 2 Change FtF (Experimental): This arm of the motivational enhancement intervention (MEI) will be delivered face to face (FtF) using a real-time, dynamic implementation approach. The intervention consisted of 2 sessions lasting approximately 60 to 90 minutes. The sessions focused on increasing participants' awareness of the multiple influences on behaviors from self, family, culture and community and how these influences impact the way we think and behave including sexually. Through a series of exercises the participant develops strategies for understanding and managing his own triggers that helps them to make healthy life choices. Both Motiv8 2Change arms used the exact same intervention, with the exception that one was delivered face to face and the other through the internet.
  Interventions: Behavioral: Entre Culturas: Navigating Culture, Identity, and HIV Risk
- Motive8 2Change -Internet (Experimental): This arm of the motivational enhancement intervention (MEI) will be delivered via the Internet face to face (FtF) using a real-time, dynamic implementation approach.The intervention consisted of 2 sessions lasting approximately 60 to 90 minutes. The sessions focused on increasing participants' awareness of the multiple influences on behaviors from self, family, culture and community and how these influences impact the way we think and behave including sexually. Through a series of exercises the participant develops strategies for understanding and managing his own triggers that helps them to make healthy life choices. Both Motiv8 2Change arms used the exact same intervention, with the exception that one was delivered face to face and the other through the internet.
  Interventions: Behavioral: Entre Culturas: Navigating Culture, Identity, and HIV Risk
- delayed (No Intervention)
- Motiv8 2Change Careers (Active Comparator): Comparable in number of sessions and duration to the experimental arms, but focused on resume development and interviewing skills. This arm consisted of 2 sessions. In the first session participants reviewed different career choices and created a winning resume. The second session focused on job interviewing skills. It included role plays with feedback. It also contains ethically mandated information regarding HIV prevention. It was delivered on line by a trained facilitator.
  Interventions: Behavioral: Entre Culturas: Navigating Culture, Identity, and HIV Risk

INTERVENTIONS:
Behavioral: Entre Culturas: Navigating Culture, Identity, and HIV Risk — A pilot test of a culturally and developmentally tailored MEI to reduce risky sex (unprotected anal sex and multiple partners) among young Hispanic men who have sex with men (YHMSM) to be delivered face-to-face (FtF) and through the Internet using a real-time implementation approach. A tailored MEI for two delivery modalities, and a health education control (HEALTH) comparable in time and number of sessions. We will test the MEI's acceptability and feasibility, obtain effect size estimates of the intervention's strength to reduce risky sex, and determine if it is ready for efficacy testing.
  Other Names: Young Hispanic MSM; HIV prevention interventions; Motiv8 2Change
  Arms: Motiv8 2Change Careers; Motive8 2 Change FtF; Motive8 2Change -Internet

SUMMARY:
The purpose of this study is to develop and pilot test a culturally and developmentally tailored Motivational Enhancement Intervention (MEI) to reduce risky sex (unprotected anal sex and multiple partners) among young Hispanic men who have sex with men (YHMSM).

DETAILED DESCRIPTION:
Stage 1, divided into Stage 1a and Stage 1b, focuses on development, refinement, and pilot testing of interventions. The formative research leading to and including intervention development is completed in Stage 1a. A pilot study to provide acceptability/feasibility data and obtain effect size estimates of the intervention's strength in changing a desired outcome is conducted in Stage 1b. If Stage 1b results are "promising," the intervention moves to full scale efficacy testing in Stage 2 using the classic experimental design of a randomized control trial (RCT). The intervention is ready for Stage 3 effectiveness testing only after its efficacy has been demonstrated in at least two Stage 2 trials.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, participants must:

1. be male;
2. self-identify as Hispanic/Latino;
3. be 18 - 29 years of age;
4. live in South Florida;
5. have had at least 1 episode of unprotected anal sex with a man in the last 6 months;
6. have had at least 2 male sex partners in the last 6 months;
7. be HIV negative or not known to be HIV positive; and
8. have not previously participated in this study.

Exclusion Criteria:

1. living with HIV infection

Ages: 18 Years to 29 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2010-08; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
The main outcome measure for the Stage 1b trial will be reduction in at least one of the two main outcome variables - number of unprotected anal sex acts and number of sex partners (both in the last 3 months). | 16 months

SECONDARY OUTCOMES:
acceptability and feasibility of the intervention | 16 months

CONTACTS AND LOCATIONS:
Overall Officials: M. Isabel Fernandez, PhD, Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University (Miami Office), Miami, Florida, United States